CLINICAL TRIAL: NCT03966066
Title: A Prospective, Multicenter Study on the Long-term Prognosis of Children With Bronchiectasis Treated With Low-dose Erythromycin
Brief Title: Long-term Prognosis of Children With Bronchiectasis Treated With Low-dose Erythromycin Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Baoping XU, Chief of Respiratory Department, Beijing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCHlung010
Record Dates: First submitted 2019-01-28; First posted 2019-05-29 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis children
MeSH Terms: conditions — Bronchiectasis | interventions — Erythromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose erythromycin group (Experimental): Erythromycin 3-5mg/kg.d orally for 6 months
  Interventions: Drug: erythromycin
- Non-erythromycin treatment group (No Intervention): systemic treatment

INTERVENTIONS:
Drug: erythromycin — 3-5mg/kg.d orally for 6 months
  Other Names: ERY
  Arms: low dose erythromycin group

SUMMARY:
According to their compliance, the children were divided into two groups: low dose erythromycin treated group (erythromycin 3-5mg/kg.d orally for 6 months) and non-erythromycin treatment group. The quality of life score and acute exacerbation were evaluated during the observation period (6 months) and one year after the withdrawal of Erythromycin.The pulmonary imaging changes and the degree of deterioration in pulmonary function were compared between the two groups.

DETAILED DESCRIPTION:
Bronchiectasis is an important chronic pulmonary disease that endangers the health of children. It is characterized by recurrent respiratory tract infection, cough, massive pus sputum, hemoptysis, etc. The chronic progression of bronchiectasis may affect the lung function of children. It affects the quality of life, growth and development, and even leads to the death of children, and brings great harm to children and their families. A New Zealand study of non-cystic fibrotic bronchiectasis found that overall forced expiratory volume at one second (FEV1) declined at an average annual rate of 1.6%. Other studies have shown a significant decline in lung function in children with bronchiectasis even after treatment. Some reports on the prognosis of children with bronchiectasis in China show that most of the children have remission in clinical symptoms, but there are still some cases of chronic recurrence and death. A non-controlled study showed that adult bronchiectasis patients who received long-term azithromycin had fewer acute exacerbations and improved symptoms, which might be associated with the antimicrobial activity and anti-inflammatory of macrolide antibiotics. In children, the effect of macrolide antibiotics on cystic fibrosis is positive. Studies have shown that macrolides can effectively improve pulmonary function and reduce the incidence of acute exacerbation of pulmonary lesions. The course of treatment is at least 6 months. For non-cystic fibrosis bronchiectasis, recent studies have shown that long-term azithromycin treatment can reduce the exacerbation of pulmonary lesions. However, the treatment of bronchiectasis children in China is still lack of standard. The aim of this study was to explore the effect of macrolides on the long term prognosis of children with bronchiectasis in China, in order to standardize the treatment and improve the prognosis of the children with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

All children participating in this clinical study must meet all of the following criteria.

1. age: 0-18 years old, male and female;
2. accord with diagnostic criteria of bronchiectasis;
3. Agreed to retain specimens related to disease research and to store them in a sample bank;
4. willing and able to cooperate with long term follow-up;
5. the guardian of the child has a good understanding of the purpose of the study, a basic understanding of the clinical research program, and voluntary participation of the child in the study and the signing of an informed consent form.

Diagnostic criteria of bronchiectasis: clinical manifestation + one or more clinical manifestations of high-resolution computed tomography (HRCT):

1. Clinical manifestations: recurrent cough, sputum, fixed wet rale in lung auscultation, clubbing finger (toe) and so on;
2. HRCT was more than one of the following: (1) In the lung segment, some distal end of a bronchial cavity diameter greater than or equal to the proximal end. the distal end of the lumen was greater than or equal to the proximal end of a segment of the bronchus. (2)The diameter of bronchus is larger than that of accompanied pulmonary artery. (3) the bronchus was seen within the area of 1.0cm under the chest wall. (4)Compared with the adjacent bronchi, the inner diameter of the bronchus was obviously larger than that of the adjacent lung segment, and the wall of the bronchus was thicker than that of the adjacent lung segment.

Exclusion Criteria:

All children with any of the following conditions must be excluded from this study:

1. children who are unable or unwilling to follow up regularly;
2. who are unable or unwilling to provide information on the history of the disease, The development of the disease and the response after treatment and other information in children.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in lung function on the spirometry | 6 months, One year after the withdrawal
  forced expiratory volume at one second (FEV1) in Liter

SECONDARY OUTCOMES:
Frequencies of pulmonary exacerbation in children | 6 months, One year after the withdrawal
  Frequencies of pulmonary exacerbation
the number of dead people | 6 months, One year after the withdrawal
  the number of people who was dead
the changes of lung image | 6 months, One year after the withdrawal
  the changes of lung image

REFERENCES:
- [Background] Pasteur MC, Bilton D, Hill AT; British Thoracic Society Bronchiectasis non-CF Guideline Group. British Thoracic Society guideline for non-CF bronchiectasis. Thorax. 2010 Jul;65 Suppl 1:i1-58. doi: 10.1136/thx.2010.136119. PMID 20627931
- [Background] Equi A, Balfour-Lynn IM, Bush A, Rosenthal M. Long term azithromycin in children with cystic fibrosis: a randomised, placebo-controlled crossover trial. Lancet. 2002 Sep 28;360(9338):978-84. doi: 10.1016/s0140-6736(02)11081-6. PMID 12383667